CLINICAL TRIAL: NCT02566616
Title: Electrical Nerve Stimulation of the Ulnar Nerve During Cubital Tunnel Decompression Surgery: Does it Improve Long Term Functional Outcomes?
Brief Title: Electrical Nerve Stimulation of the Ulnar Nerve
Acronym: ESTIM
Status: Withdrawn | Phase: Not Applicable | Type: Interventional
Why Stopped: No participants enrolled
Sponsor: University of Chicago (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 14-0646
Record Dates: First submitted 2015-09-30; First posted 2015-10-02 (Estimated); Last update posted 2017-04-05 (Actual); Status verified 2017-04

CONDITIONS: Cubital Tunnel Syndrome
MeSH Terms: conditions — Cubital Tunnel Syndrome

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Intervention (Experimental): Cubital Tunnel Release with stimulator for nerve location
  1 hour of Ulnar nerve stimulation
  Interventions: Device: Ulnar Nerve Stimulation
- Non-Intervention (Active Comparator): Cubital Tunnel Release with stimulator for nerve location NO prolonged ulnar nerve stimulation
  Interventions: Device: Ulnar Nerve Stimulation

INTERVENTIONS:
Device: Ulnar Nerve Stimulation — 1 hour of continued stimulation of the ulnar nerve using a hand held stimulator
  Other Names: Stimulation

SUMMARY:
Cubital tunnel syndrome is caused by compression of the ulnar nerve at the elbow. This leads to symptoms such as chronic hand weakness, numbness and pain. This is usually treated with a surgical procedure where the nerve is decompressed. Research has shown that nerve simulators speed up the recovery of nerves following injury. The purpose of our research is to examine the difference in patient outcomes after the nerve decompression surgery with and without nerve stimulation.

Our research questions is: What are the differences in long term functional outcomes of patients that have ulnar nerve decompression surgery with and without nerve stimulation?

DETAILED DESCRIPTION:
1. Patients will be seen in University of Chicago clinics, if they are diagnosed with Cubital Tunnel Syndrome, they will be approached to be enrolled in our study
2. If they fit inclusion and exclusion criteria, failed conservative management, and consent to be part of the study, they will be scheduled for Cubital Tunnel Surgery and randomized into intervention/non-intervention group
3. Patients will have pre-operative subjective pain and upper extremity function surveys and objective hand strength/sensation measurements done by a blinded Occupational Therapist in University of Chicago Occupational Therapy Clinic. Patient will also have a pre-operative EMG done.
4. Patient will be discharged following surgery and followed up at 6 weeks, 3 months, 6 months, 12 months. EMG will be done at 3 months and the same outcome measurements (Pain scores, PRUNE evaluation, QuickDash Questionnaire, Michigan hand Questionnaire, grip strength, sensation measurements) will be taken at each postoperative visit by the same blinded occupational therapist
5. Data will be compared pre and postoperatively

ELIGIBILITY:
Inclusion criteria

* EMG confirmed ulnar nerve neuropathy at cubital tunnel with or without these symptoms:

  * Paresthesia or numbness of the small finger and/or ring finger
  * Complaints of hand weakness
  * Exam shows positive flexion compression test at elbow and/or positive tinel's sign at the cubital tunnel
* Failed conservative management for 6 weeks

  ○ Has completed a combination of these for 6 weeks and still has symptoms
  * Night splinting in 45-60 degrees of flexion and forearm neutral
  * Padding of elbow with an elbow pad during the day
  * Daily NSAIDs if able to take them
  * Cubital tunnel steroid injection
* Age restriction: 18--65years old

Exclusion criteria

* Psychiatric conditions
* Workman's compensation patients
* Neurologic conditions (ex. MS)
* Inflammatory rheumatologic conditions (Connective tissues disease, RA… etc)
* Associated elbow and upper extremity fractures
* Previous Cubital Tunnel Surgeries
* Previous C-Spine Surgeries
* Pregnancy

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2015-11; Primary Completion 2017-04-01 (Actual); Study Completion 2017-04-01 (Actual)

PRIMARY OUTCOMES:
Patient Related Ulnar Nerve Evaluation | 10 minutes
  PRUNE Survey with 0-100 score

SECONDARY OUTCOMES:
QuickDASH | 10 minutes, pre op and each post op visit
  Survey
Michigan Hand Questionnaire | 20 minutes, pre op and each post op visit
  Survey

OTHER OUTCOMES:
EMG | Pre-op and 3 month post op visit
  Electromyelopgraph to confirm ulnar nerve neuropathy and improvement at 3 months post op
Monofilament test | 5 minutes, pre op and each post op visit
  Measure sensation on fingers
2 point discrimination | 5 minutes, pre op and each post op visit
  Measure 2 point discrimination on fingers
Pinch Strength | 5 minutes, pre op and each post op visit
  Measure Pinch strength
Grip strength | 5 minutes, pre op and each post op visit
  Measure hand grip strength

CONTACTS AND LOCATIONS:
Overall Officials: Jovito Angeles, MD, Principal Investigator — University of Chicago
Locations (1):
- University of Chicago Medical Center, Chicago, Illinois, United States